CLINICAL TRIAL: NCT00959179
Title: The Registry Evaluating Functional Outcomes of Resynchronization Management
Acronym: REFORM
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Saint Luke's Health System (Other)
Responsible Party: Dr. Brian M. Ramza, Saint Luke's Hospital
Other Study IDs: REFORM
Record Dates: First submitted 2009-08-13; First posted 2009-08-14 (Estimated); Last update posted 2009-08-14 (Estimated); Status verified 2009-08

CONDITIONS: Congestive Heart Failure
Keywords: CHF
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Device therapy patients for CHF.: enroll all consecutive patients undergoing implantable cardioverter defibrillator (ICD) and ICD with biventricular pacemaker (CRT-D) implantation for heart failure from in-patient and out-patient referral setting
- ICD and CRT-D patients: enroll all consecutive patients undergoing implantable cardioverter defibrillator (ICD) and ICD with biventricular pacemaker (CRT-D) implantation for heart failure from in-patient and out-patient referral setting

SUMMARY:
The purpose of this study is to evaluate the functional outcomes of resynchronization management and to describe the patient psychosocial characteristics (depression ad anxiety) and associated outcomes with electrophysiologic device therapy for chronic congestive heart failure.

DETAILED DESCRIPTION:
This project will prospectively enroll all consecutive patients undergoing implantable cardioverter defibrillator (ICD) and ICD with biventricular pacemaker (CRT-D) implantation for heart failure from in-patient and out-patient setting. Primary objective: Compare the psychosocial function and quality of life of ICD patients to Patients receiving CRT-D therapy. Secondary outcome objectives: 1)Determine and compare the change in LVED (left ventricular end distolic) dimension and LVESV (left ventricular end systolic volume)from baseline to 9 month follow up in CRT and ICD patient.2)Determine and compare the change in NYHA (New York Heart Association) classification, KCCQ, optimisim and pessimism, degree of stress, and social support from baseline to 9 month follow up in CRT and ICD patients. Florida Patient Acceptance Survey and Florida Shock Anxiety Scale will be determined and compared at 3 monthe and 9 months.3)Determine and compare Clinical composite score(Packer M 2002)in patient groups where: Worsened-patient dies, improved, unchanged. Inclusion Criteria: Patient referred for device therapy (ICD or CRT-D) for chronic congestive heart failure who are willing and able to give informed consent and participate in follow-up calls. Duration of patient follow up will be 9 months. Statistical Mehtodology: Univariate, Multivariatae, Kaplan-Meier analysis

ELIGIBILITY:
Inclusion Criteria:

* Patients implanted with ICD who meet Primary prevention (SCD-HeFT or MADIT II indications.
* Patients implanted with CRT-D indications (i.e. NYHA class III or IV; QRS > = to 120MS; LVEF <= TO 35%) patient willing to give informed consent and participate in follow up evaluation.

Exclusion Criteria:

* Non-English speaking patients and patients who are unable to give consent or participate in follow up protocols due to lack of a home phone or unwilling to disclose phone numbers.
* Patients with significant transient neurological impairment before, during or after device implant who have been deemed incompetent to complete the consent process, or who are unable to participate in follow-up evaluation tests.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population from In-patient and out patient setting
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2007-05; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Compare the psysocial function and quality of life of ICD patients receiving CRT with ICD therapy | 3 months and 9 month follow up

SECONDARY OUTCOMES:
Compare change in LVED&LVESV in CRT and ICD patients. Determine/compare the change in NYHA class, KCCQ, optimism/pessimism, degree of stress,social support. Florida Shock Anxiety Scale & clinical composite score determined and compared at 3 and 9 month | 9 month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Ramza, MD, Principal Investigator — Cardiovascular Consultants PA
Locations (2):
- United States (2):
  - Provena Saint Joseph Hospital, Elgin, Illinois
  - Oklahoma University Health Sciences Ctr., Oklahoma City, Oklahoma